CLINICAL TRIAL: NCT02976571
Title: Local and Intraperitoneal Analgetics in Gynecologic Laparoscopy for Post Operative Pain Relief
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0198-16-WOMC
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sub cutaneous+Intraperitoneal (Experimental): Sub cutaneous Bupivacaine+ Intraperitoneal bupivacaine
  Interventions: Drug: Bupivacaine
- Sub cutaneous+Placebo (Active Comparator): Sub cutaneous Bupivacaine+ Intraperitoneal Nacl 0.9%
  Interventions: Drug: Bupivacaine
- Placebo+Intraperitoneal (Active Comparator): Sub cutaneous Nacl 0.9%+ Intraperitoneal bupivacaine
  Interventions: Drug: Bupivacaine
- Placebo+Placebo (Placebo Comparator): Sub cutaneous Nacl 0.9%+ Intraperitoneal Nacl 0.9%
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Sub cutaneous and/or Intraperitoneal Marcaine application
  Other Names: Marcaine

SUMMARY:
A comparison between local and intraperitoneal analgetics to placebo, during laparoscopy, regarding post operative pain.

DETAILED DESCRIPTION:
4 randomly assigned groups. Grop 1 will get sub cutaneous and intraperitoneal marcain. Grop 2 will get sub cutaneous marcaine and intraperitoneal saline. Grop 3 will get sub cutaneus saline and intraperitoneal marcaine. Grop 4 will get ub cutaneous and intraperitoneal saline

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopy

Exclusion Criteria:

* Laparotomy Vaginal operations Oncologic operations Chronic use of analgetics due to pelvic pain Pregnancy Operations lasts more than 3 hours

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pain level during movement, 8 hours after laparoscopy | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Gluck, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson medical center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gluck O, Barber E, Feldstein O, Tal O, Kerner R, Keidar R, Wolfson I, Ginath S, Bar J, Sagiv R. The effect of subcutaneous and intraperitoneal anesthesia on post laparoscopic pain: a randomized controlled trial. Sci Rep. 2021 Jan 8;11(1):81. doi: 10.1038/s41598-020-80130-6. PMID 33420214